CLINICAL TRIAL: NCT06866678
Title: Can the Frailty Score Independently Predict Surgical Risk and Postoperative Morbidity in Patients With Colorectal Cancer?
Brief Title: Frailty Score and Postoperative Morbidity in Colorectal Cancer Surgery
Status: Recruiting | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Kemal ŞAHİN, M.D, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2025-02/28
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Complications; Colorectal Cancer; Frailty
MeSH Terms: conditions — Postoperative Complications; Colorectal Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail: Patients aged 65 years and older undergoing elective colorectal cancer surgery who meet three or more criteria on the Frailty Risk Index (FRI), and are classified as frail. These patients are expected to have increased vulnerability to postoperative complications.
  Interventions: Procedure: Observational Data Collection
- Non-Frail: Patients aged 65 years and older undergoing elective colorectal cancer surgery who meet fewer than three criteria on the Frailty Risk Index (FRI), and are classified as non-frail. These patients are expected to have lower risk for postoperative complications compared to the frail group.
  Interventions: Procedure: Observational Data Collection

INTERVENTIONS:
Procedure: Observational Data Collection — No intervention will be performed as part of this study. This is an observational study; all patients will receive standard perioperative care according to current clinical practice. The study will only observe and record data related to frailty status and postoperative outcomes in patients undergoing elective colorectal cancer surgery. No experimental procedures, drugs, or additional interventions will be administered.

SUMMARY:
This prospective observational study aims to evaluate the independent predictive value of the Edmonton Frailty Index (EFI) in estimating postoperative morbidity among older patients undergoing elective colorectal cancer surgery. Frailty, characterized by a decline in physiological reserves and increased vulnerability to stressors, has been recognized as a stronger predictor of adverse postoperative outcomes than chronological age alone. While the relationship between frailty and surgical outcomes has been extensively investigated in general surgical populations, data specifically focusing on patients with colorectal cancer remain limited.

In this study, patients aged 65 years and older scheduled for elective colorectal cancer surgery will undergo preoperative frailty assessment using the validated Edmonton Frailty Index (EFI). Postoperative complications, length of intensive care unit (ICU) stay, total hospital stay, and 30-day adverse outcomes, including mortality, myocardial infarction, pulmonary embolism, sepsis, and the need for reoperation, will be recorded and analyzed.

The primary objective is to determine whether frailty, as measured by the Edmonton Frailty Index, serves as an independent predictor of postoperative morbidity in this specific patient population. Secondary objectives include exploring associations between frailty and intraoperative variables such as blood loss, fluid administration, and vasopressor requirements.

By addressing this gap, the study aims to contribute to the growing body of evidence supporting the routine incorporation of frailty assessment into preoperative risk stratification protocols for older patients with colorectal cancer. The ultimate goal is to enhance perioperative risk assessment, optimize perioperative care, and improve patient outcomes.

DETAILED DESCRIPTION:
This prospective, observational study aims to evaluate whether the Frailty Risk Index (FRI) can independently predict postoperative morbidity in patients undergoing elective surgery for colorectal cancer. Frailty is a clinical syndrome characterized by decreased physiological reserve and increased vulnerability to stressors, particularly in elderly populations. Recent studies have demonstrated that frailty is a better predictor of adverse postoperative outcomes than chronological age, especially among cancer patients and the elderly surgical population.

The study will be conducted at Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital. Data will be collected from anesthesia records of patients who undergo elective colorectal cancer surgery in the General Surgery and Surgical Oncology clinics. The sample size was calculated based on the hypothesis that patients with a high Frailty Risk Score will have increased rates of postoperative morbidity. A minimum of 69 patients is required to achieve 90% power with a type I error rate of 0.05 and a medium effect size (0.5). To account for potential dropouts and missing data, a total of 80 patients will be included.

The primary objective is to assess the independent predictive value of the Frailty Risk Index for postoperative clinical outcomes in colorectal cancer patients. Secondary objectives include comparing postoperative complication rates, intensive care unit admissions, length of hospital stay, and 30-day adverse events (such as mortality, myocardial infarction, pulmonary embolism, and sepsis) between frail and non-frail patients.

Patients aged 65 years and older who are scheduled for elective colorectal cancer surgery and can be evaluated preoperatively with the FRI will be included. Exclusion criteria are emergency surgery, severe comorbidities that preclude surgery, neurological or psychiatric disorders that impair consciousness assessment, and inability or unwillingness to provide informed consent.

The Frailty Risk Index will be assessed based on five criteria: unintentional weight loss, self-reported exhaustion, weakness (reduced grip strength), slow walking speed, and low physical activity. Patients meeting three or more criteria will be classified as frail.

Data collection will include preoperative variables (age, sex, ASA score, comorbidities, diagnosis, metastasis status), intraoperative variables (anesthesia management, blood loss, fluid and blood product administration, vasopressor requirement), and postoperative outcomes (complications within 24 hours, ICU admission and stay, hospital length of stay, and adverse events within 30 days).

Statistical analysis will involve independent t-tests and chi-square tests for group comparisons, and multivariate logistic regression to assess the independent effect of the Frailty Risk Index on postoperative outcomes. A p-value of <0.05 will be considered statistically significant.

This study aims to fill a gap in the literature regarding the predictive value of frailty assessment in colorectal cancer surgery and to contribute to improved risk stratification and perioperative management in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older
* Patients undergoing surgery for colorectal cancer
* Patients scheduled for elective (non-emergency) surgery
* Individuals eligible for preoperative frailty assessment using the Edmonton Frailty Scale (EFS)
* Patients who can be followed for at least 30 days postoperatively
* Patients able to provide informed consent

Exclusion Criteria:

* Patients requiring emergency surgery
* Neurological or psychiatric disorders that prevent the assessment of consciousness level
* Severe comorbidities (Patients with extremely high surgical risk due to severe cardiovascular, respiratory, or other systemic diseases)
* Patients who do not or cannot provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective, observational study to be conducted between February 20, 2025, and June 1, 2025, in the General Surgery and Surgical Oncology departments of our hospital. The study population will consist of patients aged 18 years and older undergoing elective colorectal cancer surgery. Data will be collected from preoperative frailty assessments using the Edmonton Frailty Scale (EFS), anesthesia records, and postoperative follow-up documents
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-02 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complication Rate Postoperative Complication Rate (Clavien-Dindo ≥ Grade II) | 30 days after surgery
  The primary outcome is the incidence of postoperative complications within 30 days after surgery, classified according to the Clavien-Dindo Classification System (Grade II and above). The relationship between preoperative frailty status, measured using the Edmonton Frailty Scale (EFS), and the development of postoperative complications will be assessed.

SECONDARY OUTCOMES:
Postoperative Mortality | 30 days after surgery
  All-cause mortality within 30 days after surgery
Length of Hospital Stay | From surgery to hospital discharge (up to 30 days)
  Total length of postoperative hospital stay (in days)
ICU Admission and Length of Stay | From surgery to hospital discharge (up to 30 days)
  Requirement for ICU admission and duration of ICU stay (in days)
Surgical Site Infection | 30 days after surgery
  Incidence of surgical site infections (SSI) within 30 days after surgery
Unplanned Reoperation | 30 days after surgery
  Incidence of unplanned reoperations within 30 days after surgery
Unplanned Readmission | 30 days after discharge
  Incidence of unplanned readmission within 30 days of hospital discharge
Functional Decline | Baseline to 30 days after surgery
  Change in functional status from preoperative baseline to 30 days postoperatively
Postoperative Delirium | During hospital stay (up to 14 days)
  Incidence of postoperative delirium during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Kemal SAHIN, Principal Investigator — Ankara Oncology Education and Research Hospital Clinic of Anesthesiology and Reanimation
Locations (1):
- Dr. Abdurrahman Yurtaslan Ankara Oncology Education and Research Hospital Clinic of Anesthesiology and Rea, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmucker AM, Hupert N, Mandl LA. The Impact of Frailty on Short-Term Outcomes After Elective Hip and Knee Arthroplasty in Older Adults: A Systematic Review. Geriatr Orthop Surg Rehabil. 2019 May 6;10:2151459319835109. doi: 10.1177/2151459319835109. eCollection 2019. PMID 31105984
- [Background] Giger AW, Ditzel HM, Ewertz M, Ditzel H, Jorgensen TL, Pfeiffer P, Lund C, Ryg J. Effect of comprehensive geriatric assessment on hospitalizations in older adults with frailty initiating curatively intended oncologic treatment: The PROGNOSIS-RCT study. J Geriatr Oncol. 2024 Sep;15(7):101821. doi: 10.1016/j.jgo.2024.101821. Epub 2024 Jul 20. PMID 39034167
- [Background] Aucoin SD, Hao M, Sohi R, Shaw J, Bentov I, Walker D, McIsaac DI. Accuracy and Feasibility of Clinically Applied Frailty Instruments before Surgery: A Systematic Review and Meta-analysis. Anesthesiology. 2020 Jul;133(1):78-95. doi: 10.1097/ALN.0000000000003257. PMID 32243326
- [Background] Elsamadicy AA, Freedman IG, Koo AB, David WB, Reeves BC, Havlik J, Pennington Z, Kolb L, Shin JH, Sciubba DM. Modified-frailty index does not independently predict complications, hospital length of stay or 30-day readmission rates following posterior lumbar decompression and fusion for spondylolisthesis. Spine J. 2021 Nov;21(11):1812-1821. doi: 10.1016/j.spinee.2021.05.011. Epub 2021 May 16. PMID 34010683
- [Background] Cook MJ, Lunt M, Ashcroft DM, Board T, O'Neill TW. The impact of frailty on patient-reported outcomes following hip and knee arthroplasty. Age Ageing. 2022 Dec 5;51(12):afac288. doi: 10.1093/ageing/afac288. PMID 36571779
- [Background] Panayi AC, Orkaby AR, Sakthivel D, Endo Y, Varon D, Roh D, Orgill DP, Neppl RL, Javedan H, Bhasin S, Sinha I. Impact of frailty on outcomes in surgical patients: A systematic review and meta-analysis. Am J Surg. 2019 Aug;218(2):393-400. doi: 10.1016/j.amjsurg.2018.11.020. Epub 2018 Nov 27. PMID 30509455